CLINICAL TRIAL: NCT04595474
Title: Assessing the Prevalence of Nonalcoholic Fatty Liver Disease and Advanced Fibrosis in Patients With Type 1 Diabetes Using Vibration-Controlled Transient Elastography and Noninvasive Scores
Brief Title: Prevalence of NAFLD and Advanced Fibrosis in Patients With Type 1 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000092
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Fibrosis, Liver; Type 1 Diabetes; Cirrhosis, Liver
Keywords: Nonalcoholic fatty liver disease (NAFLD); Nonalcoholic steatohepatitis (NASH); Type 1 Diabetes; Screening; Advanced fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: 533 adult subjects with type 1 diabetes with no secondary causes of fatty liver
  Interventions: Device: Transient Elastography

INTERVENTIONS:
Device: Transient Elastography — Transient elastography is a noninvasive imaging modality used to assess NAFLD and advanced fibrosis

SUMMARY:
The aim of this study is to assess the prevalence of nonalcoholic fatty liver disease (NAFLD) in patients with type 1 diabetes receiving care at Joslin clinic using noninvasive imaging and serum-based methods with the goal of identifying high-risk patients with advanced fibrosis who should be prioritized for specialty referral

DETAILED DESCRIPTION:
This is a prospective cohort, single-center, single-arm study screening adult subjects with type 1 diabetes from the Joslin Diabetes Center outpatient clinic mainly through physician referrals for NAFLD and advanced fibrosis. Subjects will undergo a one-time screening which will last for about 30 minutes.

The following procedures will be conducted during the study visit:

1. Blood draw for metabolic measurements (HbA1c, lipid panel, ALT, AST, serum albumin, complete blood count-CBC)
2. FibroScan Measurements (LSM and CAP)
3. Anthropometric measurements (weight, height, BMI calculation, waist, and hip circumference)
4. Systolic and diastolic blood pressure

Blood Draw:

Samples of blood taken during the trial for laboratory testing will include the following metabolic measurements: AST, ALT, Platelets, percentage A1C, and lipid parameters (TC, LDL, HDL, TG).

Fibroscan: Vibration controlled transient elastography (VCTE) or FibroScan® (EchoSens, Paris, France) is a simple aid to diagnose adult patients with chronic liver diseases. FibroScan provides a fast and reliable alternative to hepatic needle biopsy. In this 5-7 minute test, the investigator induces a mild amplitude shear wave into liver tissue from a small mechanical vibrator at the end of the FibroScan probe. VCTE evaluates a representative volume of the liver that is 100-fold greater than needle biopsy and the liver stiffness measurement (LSM) is expressed in kilopascals (kPa) with values >9.8 kPa being consistent with the presence of advanced fibrosis/cirrhosis. Typically, 10 successful VCTE measurements with a median interquartile range/median ration of less than 30% are needed to have a reliable LSM.

FIB-4 Index: This is a noninvasive surrogate biomarker of advanced fibrosis that is calculated using the following formula:

FIB-4 = Age (years)×AST (U/L)/[PLT(109/L)×√ALT(U/L)] (Sterling, Lissen et al. 2006) FIB-4>2.67 is consistent with the presence of advanced fibrosis with 80% PPV.

NAFLD Fibrosis Score (NFS): This is a noninvasive surrogate biomarker of advanced fibrosis that is calculated using the following formula:

NFS= -1.675 + 0.037 - age (years) + 0.094 - BMI (kg/m2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet count (×109/l) - 0.66 × albumin (g/dl).

NFS>0.676 is consistent with the presence of advanced fibrosis

Anthropometric measurements: These include weight, height, BMI calculation, waist, and hip measurements. Measurements will be done using standardized anthropometric techniques.

Follow up may be required for High-risk patients with advanced fibrosis. If patient consents, referring or treating physicians will be notified and provided with fibroscan results for possible referral to hepatologists for further evaluation and intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female
2. Subject age between 18-75 years old
3. Subject with an established diagnosis of T1D for at least three months prior to screening

Exclusion Criteria:

1. Subject is pregnant or lactating
2. Subject has an active malignancy

4.Subject with secondary causes of fatty liver including history of any of the following:

* Hepatitis B or C virus infection
* Wilson's disease
* Lipodystrophy
* Abetalipoproteinemia
* Current or previous use of any of the following medication: amiodarone, tamoxifen, methotrexate,corticosteroids (e.g. Prednisone), or Valproate
* Male subject consuming >30 g of alcohol per day or female subject consuming >20 g of alcohol perday

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include subjects with type 1 diabetes receiving care at Joslin Diabetes Center. Addiotnal subjects from the broader Boston area may be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with NAFLD | Baseline (one time point evaluation)
  Controlled Attenuation Parameter (CAP) will be used to define the presence of NAFLD
Proportion of subjects with advanced fibrosis | Baseline (one time point evaluation)
  Transient elastography will be used to define the presence of fibrosis

SECONDARY OUTCOMES:
Proportion of subjects with advanced fibrosis per NAFLD fibrosis score-NFS | Baseline (one time point evaluation)
  NFS will be calculated using the following formula:
  NFS= -1.675 + 0.037 - age (years) + 0.094 - BMI (kg/m2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet count (×109/l) - 0.66 × albumin (g/dl).
Proportion of subjects with advanced fibrosis per Fibrosis-4 (FIB-4) index | Baseline (one time point evaluation)
  FIB-4 will be calculated using the following formula:
  FIB-4 = Age (years)×AST (U/L)/[PLT(109/L)×√ALT(U/L)]
HbA1c | Baseline (one time point evaluation)
  Association with level of diabetes control as reflected in percentage HbA1c
Anthropometrics | Baseline (one time point evaluation)
  Association with BMI and waist circumference
Lipid profile | Baseline (one time point evaluation)
  Association with lipid parameters (LDL, HDL, TG)

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, MD PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No